CLINICAL TRIAL: NCT02121548
Title: Research Project of the South Florida Center for Reducing Cancer Disparities (SUCCESS): Testing CHWs and HPV Self-Sampling to Increase Cervical Cancer Screening Among Minority Immigrants in Miami-Dade County:
Brief Title: Using CHWs and HPV Home Tests to Increase Cervical Cancer Screening in Minority Populations
Acronym: SUCCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Health Choice Network (Other); Center for Haitian Studies (Other)
Responsible Party: Principal Investigator, Olveen Carrasquillo, Chief Division of General Internal Medicine, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 20100834
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Cervical Cancer
Keywords: Screen; cervical, cancer; HPV; women; community health workers; Hispanic/ Latinas; Haitian
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Outreach (Placebo Comparator): Gets outreach materials and info on where to get screened by CHW.
  Interventions: Behavioral: CHW Outreach
- CHW Outreach (Active Comparator): Comprehensive CHW outreach including home visit, detailed 1:1 education, patient navigation
  Interventions: Behavioral: CHW Outreach and HPV Self-sampling
- CHW Outreach and HPV Self-Sampling (Active Comparator): Same as Arm 2 with a CHW outreach but also option of doing HPV home self-sampling
  Interventions: Behavioral: CHW Outreach

INTERVENTIONS:
Behavioral: CHW Outreach and HPV Self-sampling — The intervention strategies will involve three overlapping domains 1)provide health education on cervical cancer screening, 2) motivation to encourage women to have screening 3) provide navigation services to obtain the screening. We envision visits lasting no more than 60 minutes. Women who are randomized to this arm will also include information on the alternative screening method. They will be told that cervical self-sampling is an alternative screening technique for the Pap smear and they will be offered the choice of having the HPV screen done during that home visit or have a Pap Smear at the participating FQHC.
  Arms: CHW Outreach
Behavioral: CHW Outreach — The intervention strategies will involve three overlapping domains 1)provide health education on cervical cancer screening, 2) motivation to encourage women to have screening 3) provide navigation services to obtain the screening. We envision visits lasting no more than 60 minutes.
  Arms: CHW Outreach and HPV Self-Sampling; Outreach

SUMMARY:
Caribbean immigrants (both Hispanics and Blacks from Haiti) are less likely to be screened for cervical cancer than the general population. One promising approach is outreach strategies that employ Community Health Workers (CHWs). Yet even in well structured CHW programs, many women remain unscreened. In our NCI Community Networks sponsored project, we are testing an approach that combines CHWs with self sampling for the human papilloma virus (HPV) as a screening strategy among such hard to reach populations.

DETAILED DESCRIPTION:
Building on our existing community partnerships, we propose a randomized CBPR study among 600 women in three underserved communities in Miami-Dade County to determine optimal approaches to increase cervical cancer screening among Caribbean and other underserved women. The study is a three arm study with 200 women randomized at each site over 3 years. Women in the control group would be exposed to NCI approved culturally and linguistically appropriate outreach and educational materials on cervical cancer screening. Our two specific aims are 1) to determine if as compared to our control group, women randomized to the community health worker intervention group consisting one on one health education and facilitation of referrals to existing screening programs results in increase proportion of women who are screened 2) to determine if as compared to the CHW group, women randomized to a CHW intervention with the addition of a home based self-sampling strategy results in an additional increase in proportion of women who are screened versus the CHW group without HPV sampling. Secondary outcomes include comparisons of a) measures of access to care (health insurance, having a usual source of care, and visit to provider in six months) b) cost of providing the intervention in order to determine the cost of recruiting an individual woman into screening c) among women having abnormal screens, time to follow-up and further testing.

ELIGIBILITY:
Inclusion Criteria:

* Haitian, Hispanic or African American women
* ages 30-65 years
* not having had a pap smear in the last three years
* live in Miami-Dade County

Exclusion Criteria:

* having had a hysterectomy
* history of cervical cancer
* plan to move out of the neighborhood during the next six months
* are enrolled in any other cancer prevention/outreach related study

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2011-10-10 (Actual); Primary Completion 2014-07-07 (Actual); Study Completion 2015-02-17 (Actual)

PRIMARY OUTCOMES:
Having had a pap smear in last 6 months | 6 months
  Primary Outcome: The primary outcome is patient self-reporting on whether they had a Pap smear of HPV testing done since the initial evaluation. As an additional analysis, patients whom were contacted by phone but do no wish to return for follow-up evaluation will be asked by phone if they had the Pap Smear of HPV testing done.

SECONDARY OUTCOMES:
Cervical Cancer Knowledge and Access to Care | 6 months
  Cervical Cancer Knowledge: Baseline and follow-up knowledge information will also be examined as a secondary outcome.
  Access to Care: We will also examine access to care (having health insurance, usual of care of care and visits to a provider) as additional secondary outcome.

OTHER OUTCOMES:
Subgroup Analysis | 6 months
  Potential additional analysis will if the either of the two planned intervention was more efficacious among women in one location versus another. In addition using data obtained from our study questionnaire, we will also examine if there was a differential impact of the intervention among women who were uninsured, lower education, lower acculturation level or had lower levels of baseline cervical cancer knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Olveen Carrasquillo, MD, MPH, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

REFERENCES:
- [Background] Carrasquillo O, McCann S, Amofah A, Pierre L, Rodriguez B, Alonzo Y, Ilangovan K, Gonzalez M, Trevil D, Byrne MM, Koru-Sengul T, Kobetz E. Rationale and design of the research project of the South Florida Center for the Reduction of Cancer Health Disparities (SUCCESS): study protocol for a randomized controlled trial. Trials. 2014 Jul 23;15:299. doi: 10.1186/1745-6215-15-299. PMID 25056208
- [Background] Ilangovan K, Kobetz E, Koru-Sengul T, Marcus EN, Rodriguez B, Alonzo Y, Carrasquillo O. Acceptability and Feasibility of Human Papilloma Virus Self-Sampling for Cervical Cancer Screening. J Womens Health (Larchmt). 2016 Sep;25(9):944-51. doi: 10.1089/jwh.2015.5469. Epub 2016 Feb 18. PMID 26890012
- [Background] Kenya S, Okoro IS, Wallace K, Ricciardi M, Carrasquillo O, Prado G. Can Home-Based HIV Rapid Testing Reduce HIV Disparities Among African Americans in Miami? Health Promot Pract. 2016 Sep;17(5):722-30. doi: 10.1177/1524839916629970. Epub 2016 Apr 18. PMID 27091604
- [Background] Kenya S, Carrasquillo O, Fatil M, Jones J, Jean C, Huff I, Kobetz E. Human Papilloma Virus and Cervical Cancer Education Needs among HIV-Positive Haitian Women in Miami. Womens Health Issues. 2015 May-Jun;25(3):262-6. doi: 10.1016/j.whi.2014.12.007. Epub 2015 Apr 9. PMID 25864021
- [Result] Carrasquillo O, Seay J, Amofah A, Pierre L, Alonzo Y, McCann S, Gonzalez M, Trevil D, Koru-Sengul T, Kobetz E. HPV Self-Sampling for Cervical Cancer Screening Among Ethnic Minority Women in South Florida: a Randomized Trial. J Gen Intern Med. 2018 Jul;33(7):1077-1083. doi: 10.1007/s11606-018-4404-z. Epub 2018 Mar 28. PMID 29594933